CLINICAL TRIAL: NCT05714722
Title: Epiction of the Genomic and Genetic Landscape Identifies CCL5 as a Protective Factor in Colorectal Neuroendocrine Carcinoma
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, MD, Director, Zhejiang University
Other Study IDs: WFang
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Neuroendocrine Carcinomas (CRNEC); Genomic Landscape; Genetic Landscape; Prognosis; CCL5; PAX5

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Colorectal neuroendocrine carcinomas (CRNECs) are highly aggressive tumours with poor prognosis and low incidence. To date, the genomic landscape and molecular pathway alterations have not been elucidated.

Methods: Tissue sections and clinical information were collected as an in-house cohort (2010-2020). Large-scale genomic and genetic panels were applied to identify the genomic and genetic alterations of CRNEC. Through the depiction of the genomic landscape and transcriptome profile, we compared the difference between CRNEC and CR neuroendocrine tumours (CRNETs). Immunohistochemistry (IHC) staining and immunofluorescence (IF) staining were performed to confirm the genetic alterations.

ELIGIBILITY:
Inclusion Criteria:

- tissues from colorectal neuroendocrine carcinomas

Exclusion Criteria:

- no

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asia
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
overall survival | 2010-2020

SECONDARY OUTCOMES:
Comprehensive genomic and expression panels (AmoyDx® Master Panel) for dna and rna detection | 2020